CLINICAL TRIAL: NCT06383377
Title: Prospective, Multi-center, Randomized, Single Blinded and Parallel Controlled Clinical Investigation to Assess the Performance, Safety and Benefit of the Wishbone HA Medical Device, a Deproteinized Bovine Bone Material, as a Bone Graft Substitute in the Socket Management Indication Requiring Bone Grafting Procedure Before Implant Placement.
Brief Title: Evaluation of Performance, Safety and Benefit of the Wishbone HA as Bone Graft Substitute, a Pre-market Clinical Investigation
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Wishbone SA (Industry)
Collaborators: EVAMED (Other); Pharmalex (Unknown); Advimago (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Pre-market parallel study
Record Dates: First submitted 2024-04-10; First posted 2024-04-25 (Actual); Last update posted 2024-05-29 (Actual); Status verified 2024-05

CONDITIONS: Bone Regeneration; Safety Issues
MeSH Terms: interventions — Tooth Extraction; Bone Transplantation

STUDY DESIGN:
Intervention Model Description: The parallel group will be treated with the product Bio-Oss® in a 1:1 randomization. Bio- Oss® is a natural bone mineral of bovine origin. Bio-Oss® is available as granules of spongious bone. Sterilization of Bio-Oss® is carried out by irradiation. Bio-Oss® has a macro- and microporous structure similar to human spongious bone. Bio-Oss® supports the in-growth of new bone at the implantation site by serving as a stable scaffold for osteoblasts; over time it is subject to the physiological remodeling process. Bio-Oss® is slowly resorbable, depending on the physiological environment of the individual patient, or integrated into the host bone. The highly purified osteoconductive mineral structure is produced from natural bone in a multistage purification process, adhering to the strictest safety regulations.
Who Masked: Participant
Masking Description: Patients will not be informed of their randomization assignment until the 1 year post implant placement follow-up visit. At this timepoint, the primary endpoint will have been achieved (at the implant placement visit) as well as the majority of the secondary endpoints. After the bone grafting surgery, all patients will receive an identic implant cart that does not break the blinding of the study. 1 year after implant placement, the patients will receive their definitive implant cart.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Bio-Oss® (Active Comparator): Tooth scheduled for extraction will be removed in the least traumatic way. The socket will be filled with the comparator (Bio-Oss® Geistlich, granules 0.25 - 1mm). Two follow up visits to monitor the healing process will take place at 2 and 6 weeks after surgery. Implant placement will be performed 4 months after the regenerative procedure. Implant loading will be allowed after having waited a minimum of 3 months after the implant placement and after a control visit. The implant survival and success will be assessed at 3, 6 and 12 months after implant placement. A long-term follow-up will evaluate the implant survival and success at 3 and 5 years post implant placement.
  Interventions: Device: Tooth extraction and bone graft procedure
- WHA (Experimental): Tooth scheduled for extraction will be removed in the least traumatic way. The socket will be filled with the investigational device (WHA, granules 0.25- 1.0mm). Two follow up visits to monitor the healing process will take place at 2 and 6 weeks after surgery. Implant placement will be performed 4 months after the regenerative procedure. Implant loading will be allowed after having waited a minimum of 3 months after the implant placement and after a control visit. The implant survival and success will be assessed at 3, 6 and 12 months after implant placement. A long-term follow-up will evaluate the implant survival and success at 3 and 5 years post implant placement.
  Interventions: Device: Tooth extraction and bone graft procedure

INTERVENTIONS:
Device: Tooth extraction and bone graft procedure — The subject will receive a flash dose of 2 gr of amoxicillin or 600 mg of Clindamycin 1 hour before the surgery.
  Tooth will be extracted using gentle techniques to guarantee an atraumatic extraction. If the socket presents insufficient bleeding, the clinician must use an appropriate procedure to induce bleeding. The extraction site must be carefully cleaned. Extraction socket will then be filled with WHA or Bio-Oss previously hydrated with saline solution (0.9%). Extraction socket packed with the graft will be covered with a collagen sponge (Geistlich Mucograft® Seal) and sutured (cross suture, Vicryl rapide 4.0).
  If required, a limited connective tissue graft can be placed in the vestibular region.
  A CBCT scan will be performed after the bone graft procedure, i.e., after the extraction socket and the biomaterial placement, to measure the initial bone width.
  The safety of the investigational device will be evaluated.

SUMMARY:
This investigation is a pre-market, prospective, multi-center, randomized, single blinded, parallel controlled clinical investigation performed in at least 5 clinical centers for confirmatory purposes of the use of WHA as intended in the filling of extraction sockets to enhance preservation of the alveolar socket.

DETAILED DESCRIPTION:
In this study, the subjects will be pseudonymized and randomized in a 1:1 ratio between WHA and the selected comparator device Bio-Oss®. The sample size of the study has been computed based on a non-inferiority test between Bio- Oss® and WHA for device performance for the filling of extraction sockets. A total of 96 subjects will be enrolled.

The results will be used to demonstrate the safety, performance and benefit of the product WHA in the socket indication in compliance with the MDR 2017/745.

The endpoints are all accurately based on objective measurements:

* Primary Endpoint: Bone reconstruction as measured by CBCT (in mm) after bone grafting procedure.
* Secondary Endpoints:

  * Evaluation of implant stability at placement.
  * Assessment of bone density at the time of implant insertion.
  * Implant osteointegration at 3months after implant placement.
  * Evaluation of implant survival and success at 3-, 6-and12-months, 3-and 5- years after implant placement.
  * Rate of all Adverse Device Events (incidence, type, relatedness, severity, seriousness) from the time of grafting procedure up to 5 years after implant placement.
  * Patient satisfaction 6- and 12-months after implant placement.
  * Evaluation of the Sulcus index (peri-implant marginal tissue health status) at 6- and 12-months after implant placement.

ELIGIBILITY:
Inclusion Criteria:

* The subject signed the informed consent form;
* The subject is ≥ 18 and ≤ 80 years old at surgery;
* The subject is in need of a tooth extraction prior to implant placement;
* All four bony walls are preserved after extraction;
* Minimum 8mm height of bone;
* Minimum 7mm thickness of lingual vestibular;
* The subject is willing and able to comply with all investigation related procedures (such as exercising oral hygiene and attending all follow-up visits);
* Full-mouth bleeding score (FMBS) lower than 25%;
* Full-mouth plaque score (FMPI) lower than 25%.

Exclusion Criteria:

* Subject with an acute infection (abscess) at the surgical site;
* Subject with untreated periodontitis or periodontal disease;
* Subject with autoimmune diseases or subjects that had received or were currently receiving treatment with antiresorptive drugs (e.g., bisphosphonates), or steroid therapy;
* Subject who is pregnant or breastfeeding;
* Subjects is a heavy smoker (>10 cigarettes a day);
* Subject with an inability to conduct basic oral hygiene (poor oral hygiene and motivation);
* Subject with metabolic diseases (diabetes, hyperparathyroidism, osteomalacia);
* Subject with severe renal dysfunction and severe liver disease;
* Subject with known severe osteoporosis;
* Subject with multiple sclerosis and/or acromegaly;
* Subject follows radiotherapy;
* Subject with psychiatric disorders or under substance abuse (drug or alcohol);
* Subject who participates in other clinical trials interfering with the present protocol;
* Mucosal diseases in the areas to be treated.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 96 (Estimated)
Dates: Start 2024-04-26 (Actual); Primary Completion 2025-03-31 (Estimated); Study Completion 2030-03-31 (Estimated)

PRIMARY OUTCOMES:
Bone reconstruction as measured by CBCT (in mm) after bone grafting procedure. | one year
  Bone thickness will be measured using CBCT scan 4 months after the bone augmentation procedure and just before implant insertion. The most apical point from the extraction socket defined at baseline will be set as a reference. The vertical reference line will be drawn in the center of the extraction socket crossing the apical reference point. The horizontal reference line is drawn perpendicular to the vertical line crossing the apical reference point. Based on these marks, 3 measurements will be done at 1, 3 and 5 mm from the top of the crest.

SECONDARY OUTCOMES:
Assessment of the bone density at implant placement. | one year
  Assessment of the bone density on the first and second half of the defect at implant placement using a Likert scale at implant placement.
  Likert scale:
  1. = soft bone
  2. = medium bone
  3. = hard bone
Evaluation of the implant primary stability. | one year
  Implants primary stability determined by using the torque wrench at implant placement.
Assessment of the implant osteointegration after implant placement | 15 months
  Taping of the implant and a rotation test will be performed. A torque wrench will be used at 10Ncm for the rotation test.
Implant survival rate and success evaluated at 3-, 6- and 12-months and 3- and 5- To evaluate implant survival and success 3-, 6- and 12- months and 3- and 5-years after implant placement | 5 years
  At 3-, 6- and 12-months and 3- and 5-years after implant placement, implant survival will be assessed by answering if:
  1. The implant remains in the jaw.
  2. The implant is damaged to the extent that it cannot be restored.
  The success of the implant will be assessed with the criteria from Buser et al.:
  * Absence of persistent subjective complaints such as pain, foreign body sensation and/or dysesthesia
  * Absence of a peri-implant infection with suppuration
  * Absence of mobility
  * Absence of a continuous radiolucency around the implant
Collection of all adverse events (AEs) related to the device and/or procedure, and assessment of incidence, type, severity, seriousness | 5 years
  At a minimum prior and after implantation, and at each follow-up thereafter, the following treatment-emergent local AEs, namely any local AE for which the start date is on or after the date that the intervention began, will be assessed for severity, seriousness, and relatedness to the device and/or procedure and recorded in the eCRF using standard medical terminology:
  * Pain
  * Flap sloughing
  * Infection
  * Inflammation at the surgical site
  * Swelling at the surgical site
  * Bleeding
  * Bone loss
  * Loss of graft material
Evaluation of patient satisfaction at 6- and 12-months after implant placement using questionnaire. | 2 years
  The questionnaire will focus on the following questions:
  * How satisfied are you with the length of procedures and how they affected your daily functioning?
  * How satisfied are you with the function and aesthetics of the final restoration?
  * How satisfied are you with the pain associated with the treatment?
  The scale for each of these questions will be as follows:
  0= Not satisfied
  1. Fairly satisfied
  2. Satisfied
  3. Extremely satisfied
Evaluation of the peri-implant marginal tissue health status at 6 and 12 months after implant placement. | 2 years
  Assessment of the peri-implant marginal tissue health status using Sulcus Bleeding Index (mBI)
  0= No bleeding when a periodontal probe is passed along the gingival margin adjacent to the implant;
  1. Isolated bleeding spots visible;
  2. Blood forms on a confluent red line on the margin;
  3. Heavy or profuse bleeding.
Evaluation of the evolution of the interproximal bone level 3- and 12-months after implant placement. | 2 years
  The bone to implant neck distance will be evaluated at the mesial and distal aspect from the implant at 3- and 12-months post implant placement.

CONTACTS AND LOCATIONS:
Overall Officials: Bruno De Carvalho, Principal Investigator — Clinician
Locations (5):
- Belgium (5):
  - Clinique de la Source DentalMe, Louvain-la-Neuve, Brabant Wallon
  - Cabinet Debaty-Techy, Aubel, Liège
  - Clinique du Faubourg DentalMe, Chaudfontaine, Liège
  - Centre Hospitalier Université de Liège, Liège
  - Centre Oxalys, Namur

IPD SHARING:
Plan to Share IPD: Undecided